CLINICAL TRIAL: NCT01287585
Title: A Randomized, Double-Blind, Multi-Center Phase 3 Study of ADI-PEG 20 Plus Best Supportive Care (BSC) Versus Placebo Plus BSC in Subjects With Advanced Hepatocellular Carcinoma (HCC) Who Have Failed Prior Systemic Therapy
Brief Title: Ph 3 ADI-PEG 20 Versus Placebo in Subjects With Advanced Hepatocellular Carcinoma Who Have Failed Prior Systemic Therapy
Acronym: ADI-PEG 20
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Polaris Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: POLARIS2009-001
Record Dates: First submitted 2011-01-25; First posted 2011-02-01 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2016-08

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; Arginine; Arginine deiminase; ADI-PEG 20
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — ADI PEG20; Polyethylene Glycols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ADI-PEG 20 (Experimental): Arginine deiminase formulated with polyethylene glycol.
  Interventions: Drug: ADI-PEG 20 (arginine deiminase formulated with polyethylene glycol); Other: Best Supportive Care
- Placebo (Placebo Comparator): an inert treatment with no therapeutic value.
  Interventions: Drug: Placebo; Other: Best Supportive Care

INTERVENTIONS:
Drug: ADI-PEG 20 (arginine deiminase formulated with polyethylene glycol) — 18 mg/m2, weekly, intramuscular, until disease progression or toxicity.
  Arms: ADI-PEG 20
Drug: Placebo — weekly, intramuscular, until disease progression or toxicity.
  Arms: Placebo
Other: Best Supportive Care — treatment of disease-related symptoms throughout the study.

SUMMARY:
This is a study of ADI-PEG 20 (pegylated arginine deiminase), an arginine degrading enzyme versus placebo in patients with hepatocellular carcinoma who have failed prior systemic treatment (chemotherapy). Hepatocellular carcinomas have been found to require arginine, an amino acid. Thus the hypothesis is that by restricting arginine with ADI-PEG 20, the hepatocellular carcinoma cells will starve and die.

DETAILED DESCRIPTION:
Patients will be randomized 2:1 to study drug versus placebo. Patients will be recruited from North American, Europe and Asia. In addition to overall survival, progression free survival, responses by RECIST 1.1 criteria and time to tumor progression will be calculated. Safety and tolerability will be assessed, as will pharmacodynamics (peripheral blood levels of arginine and citrulline), pharmacokinetics (peripheral blood levels of ADI-PEG 20) and immunogenicity (antibodies to ADI-PEG 20).

ELIGIBILITY:
Inclusion Criteria:

* Prior diagnosis of HCC confirmed histologically.
* Prior treatment with at least 1 systemic agent, with documented progressive disease after systemic agent(s), or adverse event(s)associated with prior systemic agent(s) that resulted in discontinuance of that agent(s).
* Cirrhotic status of Child-Pugh grade B7.
* Expected survival of at least 3 months.
* Adequate hematologic, hepatic, and renal function.

Exclusion Criteria:

* Candidate for potential curative therapies (i.e., resection or transplantation) or loco-regional approaches (i.e., ablation, embolization).
* Significant cardiac disease.
* Serious infection requiring treatment with systemically administered antibiotics.
* Pregnancy or lactation.
* Expected non-compliance.
* Uncontrolled intercurrent illness, or psychiatric illness or social situations that would limit compliance with study requirements.
* Subjects who have had any anticancer treatment within 2 weeks prior to entering the study.
* Subjects who have not fully recovered from toxicities associated with previous HCC loco-regional or systemic therapies.
* Subjects with history of another primary cancer, with the exception of: a) curatively resected non-melanoma skin cancer; b) curatively treated cervical carcinoma in situ; or c) other primary solid tumor with no known active disease present in the opinion of the investigator will not affect patient outcome in the setting of current HCC diagnosis.
* Allergy to pegylated products.
* Bleeding esophageal or gastric varices within the prior three months, except if banded or treated.
* Subjects known to be HIV positive.
* Uncontrolled ascites (defined as not easily controlled with diuretic treatment).
* Having received any blood transfusion, blood component preparation, erythropoietin, albumin preparation, or granulocyte colony stimulating factors (G-CSF) within 7 days prior to screening laboratories or after screening laboratories have been obtained until first dose of study drug or placebo.
* Use of traditional medicines approved by local authorities, including but not limited to Chinese herbs within 14 days of first dose of study drug or placebo.
* ECOG performance status > 2.
* Prior allograft,including liver transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 636 (Actual)
Dates: Start 2011-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Overall survival | 18 months
  Overall survival - until death or study closure.

SECONDARY OUTCOMES:
Safety and tolerability - number of participants with adverse events. | 18 months - at anticipated end of study.
  In addition to safety and tolerability, progression free survival, response rate using RECIST 1.1 and time to tumor progression will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: John S Bomalaski, M.D., Study Director — Polaris Group
Locations (73):
- United States (21):
  - University of Alabama, Birmingham, Alabama
  - Southern California Research Center, Coronado, California
  - Catherine Frenette, La Jolla, California
  - Stanford University, Palo Alto, California
  - University of California at San Diego Moores Cancer Center, San Diego, California
  - Pacific Medical Center, San Francisco, California
  - Piedmont Research Institute, Atlanta, Georgia
  - University of Hawaii, Honolulu, Hawaii
  - University of Maryland Greenbaum Cancer Center, Baltimore, Maryland
  - Johns Hopkins University Hospital, Baltimore, Maryland
  - Wayne State University School of Medicine, Dept Oncology, Detroit, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Nebraska Hem-Onc, Lincoln, Nebraska
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Oregon, Portland, Oregon
  - Drexel University, Philadelphia, Pennsylvania
  - University of Pennsylvania Abramson Cancer Center, Philadelphia, Pennsylvania
  - UPMC Cancer Centers, Pittsburgh, Pennsylvania
  - UT Southwestern, Dallas, Texas
  - Michael E. DeBakey VA Medical Center, Houston, Texas
  - University of Washington, Seattle, Washington
- China (16):
  - A ward of Oncology-287 Changhuai Rd, Bengbu, Anhui
  - Oncology, No. 678, Furong Rd, Hefei, Anhui
  - The First Hospital of Medical University Of Anhui, Hefei, Anhui
  - 5th Fl, Inpatient Bldg, No. 8,, Fengtai Distrcit, Beijing Municipality
  - No. 156 North Road of West Second Ring, Gulou District, Fujian
  - 15th Floor, In-patient Building (East), No. 651 Dongfeng East Road, Guangzhou, Guangdong
  - 5th Fl, Inpatient Bldg, No. 71, Heti Rd, Qingxiu Disttrict, Guangxi
  - 3rd Floor, Medicine Building, No. 150 Haping Rd, Harbin, Heilongjiang
  - Oncology, 185 Road Juqian Street, Changzhou, Jiangsu
  - The Chinese people's liberation army 81 hospital, Nanjing, Jiangsu
  - 5th Floor, Medical Building, No. 1018 Huguang Rd, Changchun, Jilin
  - No. 193, Lianhe Rd, Shahekou Dist., Dalian, Liaoning
  - No. 596, Xinsi Rd., Baqiao Dist., Xi'an, Shaanxi
  - Floor 7, 3rd Inpatient Building No. 37, Guoxue Xiang, Chengdu, Sichuan
  - 13th Floor, Internal Medicine Building, No. 29 Gaotanyan Main St., Chongqing
  - Bldg No. 5, 3rd Floor, Dongan Rd, Shanghai
- Italy (10):
  - Istituto Tumori "Giovanni Paolo II", Bari
  - Policlinico S. Orsola-Malpighi, Bologna
  - Azienda Ospedaliera Niguarda Cà Granda, Milan
  - Fondazione Centro San Raffaele del Monte Tabor, Milan
  - Fondazione IRCCs "Ca Granda" Ospedale Maggiore Policlinico, Milan
  - Policlinico di Monza, Monza
  - Istituto Nazionale per lo Studio e la Cura dei Tumori, Naples
  - Azienda Ospedaliera di Padova, Padua
  - Azienda Ospedaliera San Camillo Forlanini, Roma
  - Instituto Nazionale pler le Malattie Infettive, Rome
- South Korea (5):
  - Asan Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul St. Mary's Hospital, Seoul
  - Severance Hospital, Seoul
- Taiwan (11):
  - CGMHCY, Chiayi City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Chang Gung Medical Foundation-Kaohsiung, Kaohsiung County
  - China Medicine University Hospital, Taichung
  - CMMC-LY, Tainan
  - CMMC-YK, Tainan
  - National Cheng Kung University Hospital, Tainan
  - Mackay Memorial Hospital-Taipei Branch, Taipei
  - Northern Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation-Linkou, Taoyuan
- United Kingdom (10):
  - Clatterbridge Cancer Center, Bebington
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Hammersmith Hospital, London
  - King's College Hospital, London
  - Royal Free Hospital, London
  - St. Bartholomew's Hospital, London
  - The Royal Marsden Hospital, London
  - Christie NHS Trust, Manchester
  - Nottingham University Hospital, Nottingham
  - Royal Marsden, Sutton

REFERENCES:
- [Background] Abou-Alfa GK, Qin S, Ryoo BY, Lu SN, Yen CJ, Feng YH, Lim HY, Izzo F, Colombo M, Sarker D, Bolondi L, Vaccaro G, Harris WP, Chen Z, Hubner RA, Meyer T, Sun W, Harding JJ, Hollywood EM, Ma J, Wan PJ, Ly M, Bomalaski J, Johnston A, Lin CC, Chao Y, Chen LT. Phase III randomized study of second line ADI-PEG 20 plus best supportive care versus placebo plus best supportive care in patients with advanced hepatocellular carcinoma. Ann Oncol. 2018 Jun 1;29(6):1402-1408. doi: 10.1093/annonc/mdy101. PMID 29659672